CLINICAL TRIAL: NCT04226378
Title: Canadian Real-World Outcomes of Omnipod Initiation in People With T1D: Evidence From the LMC Diabetes Registry: The COPPER Study
Brief Title: Canadian Real-World Outcomes of Omnipod Initiation in People With T1D
Acronym: COPPER
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Insulet Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: COPPER
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Observational study; Glycemic control; Insulin pumps
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Omnipod cohort: Adults with T1D who switch from MDI therapy to insulin pump therapy with Omnipod.
  Interventions: Device: Omnipod
- MDI cohort: Adults with T1D who continue MDI therapy.
  Interventions: Other: MDI

INTERVENTIONS:
Device: Omnipod — Switch from MDI therapy to an Omnipod as part of usual clinical practice. An Omnipod is a patch pump that consists of a handheld controller and a disposable pod that delivers insulin.
  Groups: Omnipod cohort
Other: MDI — Continued use of MDI therapy (traditional basal/bolus insulin regimen).
  Groups: MDI cohort

SUMMARY:
The current study aims to assess clinical outcomes in adults with type 1 diabetes (T1D) who have switched from traditional multiple daily injection (MDI) therapy to continuous subcutaneous insulin infusion (CSII) therapy with the Omnipod insulin system.

DETAILED DESCRIPTION:
Poor glycemic control is associated with increased risk of diabetes-related complications in persons with type 1 diabetes (T1D). Despite advancements in insulin therapies and an increase in diabetes technology use, only 21% of adults with T1D are meeting their targeted glycated hemoglobin (A1C) levels. The Omnipod insulin system is a patch pump that consists of a handheld controller and disposable pod that delivers insulin. A retrospective analysis of medical records in the United States found that there was a significant reduction in A1C three months after initiating Omnipod in pediatric, adolescent and adult populations with T1D who switched from either MDI or traditional CSII. Currently, the real-world effectiveness of the Omnipod compared to MDI in adults with T1D on glycemic control, weight, and insulin dose, is not established.

The Canadian Real-World Outcomes of Omnipod Initiation in People with T1D: Evidence from the LMC Diabetes Registry (COPPER) study is a retrospective, observational study using demographic and clinical data from the LMC Diabetes Registry, which consists of over 42,000 active patients with diabetes across 3 Canadian provinces. The overall objectives of this study are to assess clinical outcomes in adults with T1D who switch from MDI to CSII therapy with Omnipod, and to compare clinical outcomes in the Omnipod cohort to a matched cohort of MDI users.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T1D ≥ 12 months prior to initiating the Omnipod
* Age ≥ 18 years
* Switched from MDI to Omnipod (Omnipod cohort)
* Persistent with OmniPod treatment for ≥ six months
* No change in basal insulin type or bolus insulin type between baseline and follow up (matched MDI cohort)
* ≥ one A1C measurement during the baseline and follow-up period

Exclusion Criteria:

* Switched from traditional CSII to OmniPod
* Use of non-insulin diabetes therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with T1D initiating Omnipod between January 2011 and December 2018, and a matched cohort of MDI users who have available data during the same time frame.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (A1C) | Three to six months from baseline
  Change in A1C (%). A1C will be retrieved from the participants electronic medical records.

SECONDARY OUTCOMES:
Proportion of patients achieving A1C < 7.0% | Three to six months from baseline
  Proportion of patients achieving A1C < 7.0%
Proportion of patients achieving A1C < 8.0% | Three to six months from baseline
  Proportion of patients achieving A1C < 8.0%
Weight | Three to six months from baseline
  Change in weight (kg). Weight will be retrieved from the participants electronic medical records.
Body mass index (BMI) | Three to six months from baseline
  Change in BMI (kg/m2). BMI will be retrieved from the participants electronic medical records.
Total daily dose (TDD) of insulin | Three to six months from baseline
  Change in total daily dose (TDD) of insulin. TDD of insulin will be retrieved from the participants electronic medical records.
Weekly incidence of hypoglycemia | Three to six months from baseline
  Change in self-reported weekly incidence of any hypoglycemia. Weekly incidence of hypoglycemia will be retrieved from the participants electronic medical records.
Annual incidence of severe hypoglycemia | Three to six months from baseline
  Change in self-reported annual incidence of severe hypoglycemia. Severe hypoglycemia will be retrieved from the participants electronic medical records.

OTHER OUTCOMES:
Self-measured blood glucose (SMBG) testing frequency | Pre- and post Omnipod initiation
  The last 7 to 14 days of SMBG data during the baseline and follow-up period will be recorded from the participants electronic medical records, in a subset of participants with available SMBG data.
Change in A1C in at 12, 18, 24 and 36 months | 12 months, 18 months, 24 months and 36 months
  Change in A1C will be retrieved from the participants electronic medical records, in subsets of participants who have available A1C data at 12, 18, 24 and 36 months
Continuous glucose monitor (CGM) glucose | Three to six months from baseline
  Change in CGM glucose pre and post-Omnipod initiation will be reported in a subset of patients using a CGM device, who have 14 to 90 days of CGM data available within the baseline observation period and during the follow-up period.
CGM standard deviation (SD) | Three to six months from baseline
  Change in CGM SD pre and post-Omnipod initiation will be reported in a subset of patients using a CGM device, who have 14 to 90 days of CGM data available within the baseline observation period and during the follow-up period.
CGM Co-efficient of variation (CV) | Three to six months from baseline
  Proportion of patients with CGM CV ≤36% and >36% pre and post-Omnipod initiation will be reported in a subset of patients using a CGM device, who have 14 to 90 days of CGM data available within the baseline observation period and during the follow-up period.
Percent time in range | Three to six months from baseline
  Change in percent time in range (glucose 3.9 to 10.0 mmol/L) pre and post-Omnipod initiation will be reported in a subset of patients using a CGM device, who have 14 to 90 days of CGM data available within the baseline observation period and during the follow-up period.
Percent time below range | Three to six months from baseline
  Change in percentage time below range (glucose (<3.9 mmol/L) pre and post-Omnipod initiation will be reported in a subset of patients using a CGM device, who have 14 to 90 days of CGM data available within the baseline observation period and during the follow-up period.
Percent time above range | Three to six months from baseline
  Change in percentage time above range (glucose (>10.0 mmol/L) pre and post-Omnipod initiation will be reported in a subset of patients using a CGM device, who have 14 to 90 days of CGM data available within the baseline observation period and during the follow-up period.
A1C stratified by baseline A1C | Three to six months from baseline
  A1C outcomes will be assessed separately in patients with baseline A1C <9.0% and ≥9.0%
A1C stratified by age cohort | Three to six months from baseline
  A1C outcomes will be assessed separately in three pre-defined age cohorts: 18 to 25 years, 26 to 49 years, and ≥ 50 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, Principal Investigator — LMC Healthcare
Locations (1):
- LMC Healthcare, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brown RE, Vienneau T, Aronson R. Canadian Real-World Outcomes of Omnipod Initiation in People with Type 1 Diabetes (COPPER study): Evidence from the LMC Diabetes Registry. Diabet Med. 2021 Jun;38(6):e14420. doi: 10.1111/dme.14420. Epub 2020 Oct 22. PMID 33040383